CLINICAL TRIAL: NCT03820258
Title: A Phase 2, Open-Label, Multicenter, Multi-cohort Study to Investigate the Pharmacokinetics, Safety and Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir Fixed Dose Combination in Adolescents and Children With Chronic HCV Infection
Brief Title: Study to Investigate Pharmacokinetics, Safety and Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX) Fixed Dose Combination (FDC) in Adolescents and Children With Chronic Hepatitis C Virus (HCV) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: SOF/VEL/VOX will not be evaluated in younger age groups.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1175; 2018-000480-87 (EudraCT Number)
Record Dates: First submitted 2019-01-14; First posted 2019-01-29 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Experimental: Cohort 1 (12 to < 18 years old), 8 Weeks (Experimental): Direct-acting antiviral (DAA)-naive participants without cirrhosis in Cohort 1 (12 to < 18 years old) will receive SOF/VEL/VOX FDC 400/100/100 mg for 8 weeks.
  Interventions: Drug: SOF/VEL/VOX
- Experimental: Cohort 1 (12 to < 18 years old), 12 Weeks (Experimental): DAA-naive participants with cirrhosis or DAA-experienced participants with or without cirrhosis in Cohort 1 (12 to < 18 years old) will receive SOF/VEL/VOX FDC 400/100/100 mg for 12 weeks.
  Interventions: Drug: SOF/VEL/VOX
- Experimental: Cohort 2 (6 to < 12 years old), 8 Weeks (Experimental): DAA-naive participants without cirrhosis in Cohort 2 (6 to < 12 years old) will receive SOF/VEL/VOX FDC for 8 weeks.
  Interventions: Drug: SOF/VEL/VOX
- Experimental: Cohort 2 (6 to < 12 years old), 12 Weeks (Experimental): DAA-naive participants with cirrhosis or DAA-experienced participants with or without cirrhosis in Cohort 2 (6 to < 12 years old) will receive SOF/VEL/VOX FDC for 12 weeks.
  Interventions: Drug: SOF/VEL/VOX
- Experimental: Cohort 3 (3 to < 6 years old), 8 Weeks (Experimental): DAA-naive participants without cirrhosis in Cohort 3 (6 to < 12 years old) will receive SOF/VEL/VOX FDC for 8 weeks.
  Interventions: Drug: SOF/VEL/VOX
- Experimental: Cohort 3 (3 to < 6 years old), 12 Weeks (Experimental): DAA-naive participants with cirrhosis or DAA-experienced participants with or without cirrhosis in Cohort 3 (3 to < 6 years old) will receive SOF/VEL/VOX FDC for 12 weeks.
  Interventions: Drug: SOF/VEL/VOX

INTERVENTIONS:
Drug: SOF/VEL/VOX — Administered once daily with food.
  Other Names: Vosevi ®

SUMMARY:
The primary objective of this study is to evaluate the steady-state pharmacokinetics (PK) and confirm the age-appropriate dose of sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) fixed-dose combination (FDC) in pediatric participants with chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
Participants will receive placebo to match SOF/VEL/VOX FDC to assess ability to swallow tablets at screening up to Day 1.

ELIGIBILITY:
Key Inclusion Criteria:

* Consent of parent or legal guardian required
* Chronic HCV infection
* Screening laboratory values within defined thresholds
* Individuals must have a determination of prior treatment status:

  * DAA-naive is defined as either:

    * Treatment naive with no prior exposure to any interferon (IFN), ribavirin (RBV), or approved or experimental HCV-specific DAA
    * Treatment experienced with an IFN-based regimen and no prior exposure to an approved or experimental HCV-specific DAA
  * DAA-experienced is defined as prior exposure to a regimen including any DAA (eg, non-structural protein (NS)3/4A protease inhibitor, NS5A inhibitor, or NS5B nucleotide/nucleoside inhibitor)

Key Exclusion Criteria:

* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Co-infection with human immunodeficiency virus (HIV), acute hepatitis A virus (HAV) or hepatitis B virus (HBV)
* Clinical hepatic decompensation (eg, clinical ascites, encephalopathy, and/or variceal hemorrhage)
* Pregnant or nursing females
* Known hypersensitivity to study medication
* Use of any prohibited concomitant medications as within 28 days of the Day 1 visit

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (10):
- Italy (5):
  - SOS-intraSOC Epatologia, Florence
  - Servizio di Epatologia e Nutrizione Pediatrica, Milan
  - US Infettivologia Pediatrica-Polo Universitario, Milan
  - UOS Epatologia Pediatrica, Napoli
  - UOSD Epatologia, San Giovanni Rotondo
- Poland (3):
  - Wojewodzki Szpital, Bydgoszcz
  - Med Polonia, Poznan
  - Uniwersytecki Szpital Kliniczny im., Wroclaw
- United Kingdom (2):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Kings Healthcare NHS Trust Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe. The first participant was screened on 28 January 2019. The last study visit occurred on 19 February 2020.
Pre-assignment Details: The study was terminated because EMA granted Gilead a waiver for SOF/VEL/VOX in children less than 12 years old. Cohorts 2 and 3 were not enrolled. As per the protocol, participants could have received 8 or 12 weeks of treatment, depending on their prior treatment and disease status, however all participants received treatment for 8 weeks.
Groups:
- SOF/VEL/VOX FDC: Direct-acting antiviral (DAA) - naive participants without cirrhosis (12 to < 18 years old) received sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) fixed-dose (FDC) combination (400/100/100 mg tablet) orally once daily in nonfasting state for 8 weeks. A single placebo to match tablet was administered during screening until Day 1 to confirm the participant was able to swallow SOF/VEL/VOX 400/100/100 mg tablets.
Period: Overall Study
Arm/Group | SOF/VEL/VOX FDC
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 16
  Race: Black or African American | 1
  Race: Asian | 2
  Race: Other | 2
  Race: American Indian or Alaska Native | 0
  Race: Native Hawaiian or Pacific Islander | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 13
  Poland | 4
  United Kingdom | 4
Cirrhosis [Count of Participants; unit: Participants]
  Yes | 0
  No | 21
Baseline HCV Ribonucleic acid (RNA) [Mean (Standard Deviation); unit: log10 IU/mL] | 5.9 (0.70)
Baseline Alanine aminotransferase (ALT) Category [Count of Participants; unit: Participants]
  ≤ 1.5 x (Upper Limit of Normal) ULN | 16
  > 1.5 x ULN | 5

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of SOF, GS-331007 (Metabolite of SOF), VEL, and VOX
Description: AUCtau was defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval). For participants with separate consent to participate in the optional intensive PK substudy, intensive serial PK blood samples were collected at Week 2 or Week 4. Sparse PK samples were collected from all participants at Weeks 1, 2, 4, and end of treatment/Week 8. Plasma concentration data from all PK samples (intensive and sparse) were combined and used to generate PK parameters of SOF, GS-331007, VEL, and VOX for all participants using a population PK modeling approach.
Time Frame: Sparse PK Sample (all participants): At Weeks 1 and 8 at any time, Weeks 2 and 4 (predose and between 15 minutes and 4 hours postdose). Intensive PK Sample [PK Substudy (N=14)]: Week 2 or Week 4 (0 (predose), 0.5, 1, 2, 3, 4, 6, 8, and 12 hours postdose)
Population: The Pharmacokinetic Analysis Set included all enrolled adolescent participants who received at least 1 dose of study drug and for whom at least 1 nonmissing PK concentration value was available from all types of PK sampling.
Measure: Mean (Standard Deviation); unit: hours•nanogram/milliliter
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
hours•nanogram/milliliter
  SOF | 2474.8 (1247.28)
  GS- 331007 (metabolite of SOF) | 14890.2 (3126.35)
  VEL | 6773.0 (2367.30)
  VOX | 2205.8 (1403.45)

2. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug Due to an Adverse Event
Description: Treatment-emergent Adverse Events (TEAE) were defined as events that met 1 or both of the following criteria as any AEs with onset dates on or after the study drug start date and no later than 30 days after the permanent discontinuation of study drug. It also includes the AEs that leads to premature discontinuation of study drug.
Time Frame: First dose date up to the last dose date (maximum: 8 Weeks) plus 30 days
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR was defined as hepatitis C virus (HCV RNA) < Lower limit of quantification (LLOQ) (ie, < 15 IU/mL) 12 weeks after discontinuation of the study drug.
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set included all adolescent participants 12 to < 18 years old who were enrolled into the study and took at least 1 dose of study drug (SOF/VEL/VOX FDC).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 100.0 [83.9 to 100.0]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR was defined as HCV RNA < LLOQ (ie, < 15 IU/mL) 4 weeks after discontinuation of the study drug.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 100.0 [83.9 to 100.0]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR was defined as HCV RNA < LLOQ (ie, < 15 IU/mL) 24 weeks after discontinuation of the study drug.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 100.0 [83.9 to 100.0]

6. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Overall Virologic Failure comprises of on-treatment virologic failure and relapse. On-treatment virologic failure (breakthrough, rebound, and nonresponse) and relapse were defined as follows: Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), Rebound (confirmed > 1 log10IU/mL increase in HCV RNA from nadir while on treatment), or Nonresponse (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment) and Relapse (confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on treatment visit).
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 0

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Description: Percentage of participants with HCV RNA < LLOQ (15 IU/mL) while on treatment by analysis visit.
Time Frame: Weeks 1, 2, 4, and 8
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants
  Week 1 | 52.4 [29.8 to 74.3]
  Week 2 | 81.0 [58.1 to 94.6]
  Week 4 | 90.5 [69.6 to 98.8]
  Week 8 | 100.0 [83.9 to 100.0]

8. Secondary Outcome: Percentage of Participants Who Developed Viral Resistance to SOF, VEL, and/or VOX During Treatment
Description: Plasma samples were collected and stored for potential HCV sequencing. Impact on the treatment outcomes of SVR12 and SVR24 were observed during the study. Baseline nonstructural protein (NS)3, NS5A, and NS5B deep sequencing analysis was performed for all participants. Sequencing for the HCV NS5A and NS5B regions was performed for all enrolled participants at baseline and for participants with virologic failure.
Time Frame: Up to End of Treatment (Week 8)
Population: Resistance Analysis Population was defined as all participants in the Safety Analysis Set with a virologic outcome. No on-treatment virologic breakthrough or relapse was observed. Therefore, no participants qualified for resistance testing.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 0

9. Secondary Outcome: Percentage of Participants Who Developed Viral Resistance to SOF, VEL, and/or VOX When Treatment is Discontinued
Description: as for outcome 8
Time Frame: Up to Posttreatment Week 24
Population: Resistance Analysis Population was defined as all participants in the Safety Analysis Set with a virologic outcome. No on-treatment virologic breakthrough or relapse was observed through posttreatment Week 12 or posttreatment Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants | 0

10. Secondary Outcome: Change in HCV RNA From Day 1 Through End of Treatment
Time Frame: Baseline (Day 1); Weeks 1, 2 ,4, and 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
log10 IU/mL
  Change at Week 1: number analyzed (Participants) | 20
  Change at Week 1 | -4.55 (0.525)
  Change at Week 2 | -4.65 (0.621)
  Change at Week 4: number analyzed (Participants) | 20
  Change at Week 4 | -4.71 (0.661)
  Change at Week 8 | -4.77 (0.698)

11. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization
Description: ALT normalization was defined as ALT > upper limit of normal (ULN) at baseline and ALT ≤ ULN at each visit.
Time Frame: Baseline (Day 1); Week 1, 2, 4, 8, and Posttreatment/Follow-up Week 4 (FU-4)
Population: Participants in the Full Analysis Set with available data were analyzed. It includes participants with ALT >ULN at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 5
percentage of participants
  Week 1: number analyzed (Participants) | 4
  Week 1 | 50.0
  Week 2: number analyzed (Participants) | 4
  Week 2 | 75.0
  Week 4 | 100.0
  Week 8 | 100.0
  FU-4: number analyzed (Participants) | 4
  FU-4 | 100.0

12. Secondary Outcome: Change From Baseline in Height Percentiles as a Measurement of Growth and Development
Description: An age- and sex-specific percentile was derived for each weight, height, and body mass index (BMI) measurement according to the statistical analysis system (SAS) program available on the Centers for Disease Control and Prevention (CDC) website using the year 2000 growth charts.
Time Frame: Baseline (Day 1); Weeks 1, 2, 4, 8, FU-4, Posttreatment/Follow-up Week 12 (FU-12), and Posttreatment/Follow-up Week 24 (FU-24)
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentile
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentile
  Baseline | 47.9 [32.4 to 63.2]
  Change at Week 8 | 0.0 [-3.0 to 1.3]
  Change at FU-12 | 0.0 [-2.2 to 3.8]
  Change at FU-24 | -0.2 [-3.1 to 4.3]

13. Secondary Outcome: Change From Baseline in Weight Percentiles as a Measurement of Growth and Development
Description: as for outcome 12
Time Frame: Baseline (Day 1); Weeks 1, 2, 4, 8, FU-4, FU-12, and FU-24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentile
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentile
  Baseline | 54.0 [30.9 to 75.9]
  Change at Week 8 | -2.5 [-3.5 to -1.2]
  Change at FU-12 | -2.7 [-7.1 to 0.3]
  Change at FU-24 | -1.6 [-5.2 to 4.3]

14. Secondary Outcome: Number of Participants by Tanner Stage Assessment as a Measurement of Growth and Development
Description: Tanner Pubertal Staging were assessed for pubic hair growth and genitalia development (males) and for pubic hair growth and breast development (females) in stages 1 to 5. Tanner stages will be used to evaluate the onset and progression of pubertal changes from stage 1 (pre-pubertal) to stage 5 (adult). If a participant had reached Tanner stage 5, no further Tanner pubertal stage assessments were to be completed.Pubic hair growth: Tanner stages (1: No hair, 2: Downy hair, 3: More coarse and curly hair, 4: Adult-like hair quality; 5: Hair extends to medial surface of the thighs); Breast development: Tanner stages (1: No glandular tissue, 2: Breast bud forms,3: More elevated, outside areola, 4: Increased breast size,5: Final adult-size breasts); Genitalia development: Tanner stages (1: Testes, scrotum, and penis about same size, 2: Enlargement of scrotum and testes, Penis (10.5-12.5); 3: Enlargement of penis (11.5-14); 4: Penis size (13.5-15); 5: Genitalia adult in size and shape).
Time Frame: Baseline (Day 1); Weeks 8, FU-12, and FU-24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
Participants
  Pubic Hair (Male); Baseline: number analyzed (Participants) | 8
  Pubic Hair (Male); Baseline: Stage 1 | 1
  Pubic Hair (Male); Baseline: Stage 2 | 1
  Pubic Hair (Male); Baseline: Stage 3 | 0
  Pubic Hair (Male); Baseline: Stage 4 | 4
  Pubic Hair (Male); Baseline: Stage 5 | 2
  Pubic Hair (Male); Week 8: number analyzed (Participants) | 8
  Pubic Hair (Male); Week 8: Stage 1 | 0
  Pubic Hair (Male); Week 8: Stage 2 | 2
  Pubic Hair (Male); Week 8: Stage 3 | 0
  Pubic Hair (Male); Week 8: Stage 4 | 4
  Pubic Hair (Male); Week 8: Stage 5 | 2
  Pubic Hair (Male); FU-12: number analyzed (Participants) | 8
  Pubic Hair (Male); FU-12: Stage 1 | 0
  Pubic Hair (Male); FU-12: Stage 2 | 2
  Pubic Hair (Male); FU-12: Stage 3 | 0
  Pubic Hair (Male); FU-12: Stage 4 | 3
  Pubic Hair (Male); FU-12: Stage 5 | 3
  Pubic Hair (Male); FU-24: number analyzed (Participants) | 8
  Pubic Hair (Male); FU-24: Stage 1 | 0
  Pubic Hair (Male); FU-24: Stage 2 | 1
  Pubic Hair (Male); FU-24: Stage 3 | 1
  Pubic Hair (Male); FU-24: Stage 4 | 2
  Pubic Hair (Male); FU-24: Stage 5 | 4
  Genitalia (Male); Baseline: number analyzed (Participants) | 8
  Genitalia (Male); Baseline: Stage 1 | 1
  Genitalia (Male); Baseline: Stage 2 | 1
  Genitalia (Male); Baseline: Stage 3 | 0
  Genitalia (Male); Baseline: Stage 4 | 4
  Genitalia (Male); Baseline: Stage 5 | 2
  Genitalia (Male); Week 8: number analyzed (Participants) | 8
  Genitalia (Male); Week 8: Stage 1 | 0
  Genitalia (Male); Week 8: Stage 2 | 2
  Genitalia (Male); Week 8: Stage 3 | 0
  Genitalia (Male); Week 8: Stage 4 | 4
  Genitalia (Male); Week 8: Stage 5 | 2
  Genitalia (Male); FU-12: number analyzed (Participants) | 8
  Genitalia (Male); FU-12: Stage 1 | 0
  Genitalia (Male); FU-12: Stage 2 | 2
  Genitalia (Male); FU-12: Stage 3 | 0
  Genitalia (Male); FU-12: Stage 4 | 3
  Genitalia (Male); FU-12: Stage 5 | 3
  Genitalia (Male); FU-24: number analyzed (Participants) | 8
  Genitalia (Male); FU-24: Stage 1 | 0
  Genitalia (Male); FU-24: Stage 2 | 1
  Genitalia (Male); FU-24: Stage 3 | 1
  Genitalia (Male); FU-24: Stage 4 | 2
  Genitalia (Male); FU-24: Stage 5 | 4
  Pubic Hair (Female); Baseline: number analyzed (Participants) | 13
  Pubic Hair (Female); Baseline: Stage 1 | 0
  Pubic Hair (Female); Baseline: Stage 2 | 2
  Pubic Hair (Female); Baseline: Stage 3 | 2
  Pubic Hair (Female); Baseline: Stage 4 | 5
  Pubic Hair (Female); Baseline: Stage 5 | 4
  Pubic Hair (Female); Week 8: number analyzed (Participants) | 13
  Pubic Hair (Female); Week 8: Stage 1 | 0
  Pubic Hair (Female); Week 8: Stage 2 | 2
  Pubic Hair (Female); Week 8: Stage 3 | 1
  Pubic Hair (Female); Week 8: Stage 4 | 5
  Pubic Hair (Female); Week 8: Stage 5 | 5
  Pubic Hair (Female); FU-12: number analyzed (Participants) | 13
  Pubic Hair (Female); FU-12: Stage 1 | 0
  Pubic Hair (Female); FU-12: Stage 2 | 2
  Pubic Hair (Female); FU-12: Stage 3 | 1
  Pubic Hair (Female); FU-12: Stage 4 | 5
  Pubic Hair (Female); FU-12: Stage 5 | 5
  Pubic Hair (Female); FU-24: number analyzed (Participants) | 13
  Pubic Hair (Female); FU-24: Stage 1 | 0
  Pubic Hair (Female); FU-24: Stage 2 | 1
  Pubic Hair (Female); FU-24: Stage 3 | 2
  Pubic Hair (Female); FU-24: Stage 4 | 4
  Pubic Hair (Female); FU-24: Stage 5 | 6
  Breasts (Female); Baseline: number analyzed (Participants) | 13
  Breasts (Female); Baseline: Stage 1 | 0
  Breasts (Female); Baseline: Stage 2 | 2
  Breasts (Female); Baseline: Stage 3 | 2
  Breasts (Female); Baseline: Stage 4 | 4
  Breasts (Female); Baseline: Stage 5 | 5
  Breasts (Female); Week 8: number analyzed (Participants) | 13
  Breasts (Female); Week 8: Stage 1 | 0
  Breasts (Female); Week 8: Stage 2 | 2
  Breasts (Female); Week 8: Stage 3 | 1
  Breasts (Female); Week 8: Stage 4 | 5
  Breasts (Female); Week 8: Stage 5 | 5
  Breasts (Female); FU-12: number analyzed (Participants) | 13
  Breasts (Female); FU-12: Stage 1 | 0
  Breasts (Female); FU-12: Stage 2 | 2
  Breasts (Female); FU-12: Stage 3 | 1
  Breasts (Female); FU-12: Stage 4 | 5
  Breasts (Female); FU-12: Stage 5 | 5
  Breasts (Female); FU-24: number analyzed (Participants) | 13
  Breasts (Female); FU-24: Stage 1 | 0
  Breasts (Female); FU-24: Stage 2 | 1
  Breasts (Female); FU-24: Stage 3 | 2
  Breasts (Female); FU-24: Stage 4 | 4
  Breasts (Female); FU-24: Stage 5 | 6

15. Secondary Outcome: Change From Baseline in Radiographic Bone Age Assessment as a Measurement of Growth and Development
Description: For radiographic bone age assessment, a single x-ray of the left wrist, hand, and fingers was performed and assessed by changes from baseline through end of treatment period.
Time Frame: Baseline (Day 1); Week 8
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
years
  Baseline | 14.5 [13.7 to 16.0]
  Change at Week 8 | 0.0 [0.0 to 0.5]

16. Secondary Outcome: Change From Baseline in C-Type Collagen Sequence (CTX) Bone Turn-Over Biochemical Marker as a Measurement of Growth and Development
Description: Fasting blood samples for baseline values for bone age biomarkers CTX and change from baseline were recorded.
Time Frame: Baseline (Day 1); FU-24
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
ng/mL
  Baseline | 1.35 [1.05 to 2.35]
  Change at FU-24 | -0.22 [-0.55 to -0.04]

17. Secondary Outcome: Change From Baseline in Procollagen Type 1 N-Terminal Propeptide (P1NP) Bone Turn-Over Biochemical Marker as a Measurement of Growth and Development
Description: Fasting blood samples for baseline values for bone age biomarkers P1NP and change from baseline were recorded.
Time Frame: Baseline (Day 1); FU-24
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 20
ng/mL
  Baseline | 383.25 [175.00 to 944.20]
  Change at FU-24 | -101.50 [-359.00 to -24.98]

18. Secondary Outcome: Percentage of Participants in Each Swallowability Category of Able to Swallow or Unable to Swallow SOF/VEL/VOX 400/100/100 mg Size Tablets
Description: Swallowability for SOF/VEL/VOX FDC placebo to match (PTM) tablets was summarized based on the participants present in each swallowability category of Able to Swallow or Unable to Swallow a placebo tablet on one occasion during screening until Day 1.
Time Frame: Baseline (Day 1)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants
  Able to Swallow PTM Tablet | 100.0
  Unable to Swallow PTM Tablet | 0

19. Secondary Outcome: Percentage of Participants With Acceptability Questionnaire Responses as Assessed by the Study Participant
Description: A questionnaire was administered to participants to assess acceptability, including palatability, of the formulation. Acceptability and palatability were assessed by questions about how the study drug tasted, how easy it was to swallow the study drug, and also at the end of treatment about how it was to take the study drug and, as they all received a single tablet daily, how they felt about the number of tablets they had to swallow.
Time Frame: Baseline (Day 1); Week 8
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants
  Did Not Taste Study Drug; Day 1 | 23.8
  Taste (Very Bad); Day 1 | 9.5
  Taste (Bad); Day 1 | 9.5
  Taste (Maybe Bad/ Maybe Good); Day 1 | 38.1
  Taste (Good); Day 1 | 19.0
  Taste (Very Good); Day 1 | 0
  Swallow (Very Hard); Day 1 | 9.5
  Swallow (Hard); Day 1 | 9.5
  Swallow (Maybe Hard/ Maybe Easy); Day 1 | 9.5
  Swallow (Easy); Day 1 | 23.8
  Swallow (Very Easy); Day 1 | 47.6
  Did Not Taste Study Drug; Week 8: number analyzed (Participants) | 20
  Did Not Taste Study Drug; Week 8 | 25.0
  Taste (Very Bad); Week 8: number analyzed (Participants) | 20
  Taste (Very Bad); Week 8 | 0
  Taste (Bad); Week 8: number analyzed (Participants) | 20
  Taste (Bad); Week 8 | 25.0
  Taste (Maybe Bad/ Maybe Good); Week 8: number analyzed (Participants) | 20
  Taste (Maybe Bad/ Maybe Good); Week 8 | 40.0
  Taste (Good); Week 8: number analyzed (Participants) | 20
  Taste (Good); Week 8 | 5.0
  Taste (Very Good); Week 8: number analyzed (Participants) | 20
  Taste (Very Good); Week 8 | 5.0
  Swallow (Very Hard); Week 8: number analyzed (Participants) | 20
  Swallow (Very Hard); Week 8 | 0
  Swallow (Hard); Week 8: number analyzed (Participants) | 20
  Swallow (Hard); Week 8 | 5.0
  Swallow (Maybe Hard/ Maybe Easy); Week 8: number analyzed (Participants) | 20
  Swallow (Maybe Hard/ Maybe Easy); Week 8 | 20.0
  Swallow (Easy); Week 8: number analyzed (Participants) | 20
  Swallow (Easy); Week 8 | 25.0
  Swallow (Very Easy); Week 8: number analyzed (Participants) | 20
  Swallow (Very Easy); Week 8 | 50.0
  Take (Very Hard); Week 8: number analyzed (Participants) | 20
  Take (Very Hard); Week 8 | 0
  Take (Hard); Week 8: number analyzed (Participants) | 20
  Take (Hard); Week 8 | 0
  Take (Maybe Hard/Maybe Easy); Week 8: number analyzed (Participants) | 20
  Take (Maybe Hard/Maybe Easy); Week 8 | 25.0
  Take (Easy); Week 8: number analyzed (Participants) | 20
  Take (Easy); Week 8 | 50.0
  Take (Very Easy); Week 8: number analyzed (Participants) | 20
  Take (Very Easy); Week 8 | 25.0
  Number of Tablets(Very Hard); Week 8: number analyzed (Participants) | 20
  Number of Tablets(Very Hard); Week 8 | 0
  Number of Tablets(Hard); Week 8: number analyzed (Participants) | 20
  Number of Tablets(Hard); Week 8 | 0
  Number of Tablets( Maybe Hard/ Maybe Easy); Week 8: number analyzed (Participants) | 20
  Number of Tablets( Maybe Hard/ Maybe Easy); Week 8 | 45.0
  Number of Tablets(Easy); Week 8: number analyzed (Participants) | 20
  Number of Tablets(Easy); Week 8 | 25.0
  Number of Tablets(Very Easy); Week 8: number analyzed (Participants) | 20
  Number of Tablets(Very Easy); Week 8 | 30.0

20. Secondary Outcome: Percentage of Participants With Acceptability Questionnaire Responses as Assessed by the Parent/Legal Guardian
Description: A questionnaire was administered to the parent/legal guardian of participants to assess acceptability, including palatability, of the formulation. Acceptability and palatability were assessed by questions about how the study drug tasted, how easy it was to swallow the study drug, about how it was to take the study drug and, as they all received a single tablet daily, how they felt about the number of tablets they had to swallow.
Time Frame: Week 8
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
percentage of participants
  Did Not Taste Study Drug | 61.9
  Taste (Very Bad) | 0
  Taste (Bad) | 23.8
  Taste (Maybe Bad/ Maybe Good) | 9.5
  Taste (Good) | 4.8
  Taste (Very Good) | 0
  Swallow (Very Hard) | 4.8
  Swallow (Hard) | 9.5
  Swallow (Maybe Hard/ Maybe Easy) | 14.3
  Swallow (Easy) | 33.3
  Swallow (Very Easy) | 38.1
  Take (Very Hard) | 0
  Take (Hard) | 9.5
  Take (Maybe Hard/ Maybe Easy) | 19.0
  Take (Easy) | 47.6
  Take (Very Easy) | 23.8
  Number of Tablets (Very Hard) | 0
  Number of Tablets (Hard) | 4.8
  Number of Tablets (Maybe Hard/Maybe Easy) | 28.6
  Number of Tablets (Easy) | 47.6
  Number of Tablets (Very Easy) | 19.0

21. Secondary Outcome: Neuropsychiatric Assessments Based on Questionnaire as Completed by Participant
Description: Neuropsychiatric safety assessment was done using the Pediatric Quality of Life (PedsQL™ 4.0 SF15). The PedsQL™ 4.0 SF15 Questionnaires was completed by all participants. It is a comprehensive and widely used patient-reported outcome survey designed to measure health-related quality of life in healthy children and adolescents. It is presented for each of the 4 domains of the SF-15 (physical functioning, emotional functioning, social functioning, and school functioning), the psychosocial health summary (emotional, social, and school functioning domains), physical health summary and the Total Score. Total scores as well as each of the subscale scores are transformed on a scale from 0 to 100. Higher scores in each case indicate better health-related quality of life (HRQOL). A positive change from end of treatment period indicates improvement.
Time Frame: Weeks 8, FU-12, and FU-24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
score on a scale
  Physical Functioning; Week 8 | 88.1 (17.06)
  Physical Functioning; Change at FU-12 | -0.7 (7.29)
  Physical Functioning; Change at FU-24 | -0.9 (6.40)
  Emotional Functioning; Week 8 | 78.0 (19.33)
  Emotional Functioning; Change at FU-12 | -3.0 (21.43)
  Emotional Functioning; Change at FU-24 | -1.8 (18.56)
  Social Functioning; Week 8: number analyzed (Participants) | 20
  Social Functioning; Week 8 | 95.0 (10.95)
  Social Functioning; Change at FU-12: number analyzed (Participants) | 20
  Social Functioning; Change at FU-12 | -2.9 (8.67)
  Social Functioning; Change at FU-24: number analyzed (Participants) | 20
  Social Functioning; Change at FU-24 | -0.4 (6.88)
  School Functioning; Week 8 | 80.2 (22.89)
  School Functioning; Change at FU-12 | -4.8 (18.37)
  School Functioning; Change at FU-24 | -3.6 (16.15)
  Physical Health; Week 8 | 88.1 (17.06)
  Physical Health ; Change at FU-12 | -0.7 (7.29)
  Physical Health; Change at FU-24 | -0.9 (6.40)
  Psychosocial Health; Week 8 | 83.6 (15.04)
  Psychosocial Health; Change at FU-12 | -3.6 (12.38)
  Psychosocial Health; Change at FU-24 | -2.4 (11.51)
  Total Score; Week 8 | 85.1 (14.13)
  Total Score; Change at FU-12 | -2.6 (9.32)
  Total Score; Change at FU-24 | -1.9 (8.83)

22. Secondary Outcome: Neuropsychiatric Assessments Based on Questionnaire as Completed by Parent/Legal Guardian
Description: Neuropsychiatric safety assessment was done using the Pediatric Quality of Life (PedsQL™ 4.0 SF15). The PedsQL™ 4.0 SF15 Questionnaires was completed by the parent/ legal guardian of the participants. It is a comprehensive and widely used patient-reported outcome survey designed to measure health-related quality of life in healthy children and adolescents. It is presented for each of the 4 domains of the SF-15 (physical functioning, emotional functioning, social functioning, and school functioning), the psychosocial health summary (emotional, social, and school functioning domains), physical health summary and the Total Score. Total scores as well as each of the subscale scores are transformed on a scale from 0 to 100. Higher scores in each case indicate better HRQOL. A positive change from end of treatment period indicates improvement.
Time Frame: Weeks 8, FU-12, and FU-24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
score on a scale
  Physical Functioning; Week 8 | 87.4 (17.29)
  Physical Functioning; Change at FU-12: number analyzed (Participants) | 20
  Physical Functioning; Change at FU-12 | -2.5 (9.39)
  Physical Functioning; Change at FU-24 | -1.7 (12.97)
  Emotional Functioning; Week 8 | 78.6 (21.06)
  Emotional Functioning; Change at FU-12: number analyzed (Participants) | 20
  Emotional Functioning; Change at FU-12 | -0.3 (22.53)
  Emotional Functioning; Change at FU-24 | -2.4 (17.95)
  Social Functioning; Week 8 | 87.7 (17.80)
  Social Functioning; Change at FU-12: number analyzed (Participants) | 20
  Social Functioning; Change at FU-12 | 4.2 (18.04)
  Social Functioning; Change at FU-24 | 0.8 (14.41)
  School Functioning; Week 8 | 74.2 (27.63)
  School Functioning; Change at FU-12: number analyzed (Participants) | 20
  School Functioning; Change at FU-12 | 3.3 (20.84)
  School Functioning; Change at FU-24 | 3.2 (16.77)
  Physical Health; Week 8 | 87.4 (17.29)
  Physical Health ; Change at FU-12: number analyzed (Participants) | 20
  Physical Health ; Change at FU-12 | -2.5 (9.39)
  Physical Health; Change at FU-24 | -1.7 (12.97)
  Psychosocial Health; Week 8 | 80.0 (17.46)
  Psychosocial Health; Change at FU-12: number analyzed (Participants) | 20
  Psychosocial Health; Change at FU-12 | 2.1 (15.82)
  Psychosocial Health; Change at FU-24 | 0.2 (9.61)
  Total Score; Week 8 | 82.5 (16.10)
  Total Score; Change at FU-12: number analyzed (Participants) | 20
  Total Score; Change at FU-12 | 0.6 (12.67)
  Total Score; Change at FU-24 | -0.4 (7.87)

23. Secondary Outcome: Change From Baseline in Neuropsychiatric Assessments as Completed by Participant
Description: Neuropsychiatric safety assessment was done using the Pediatric Quality of Life (PedsQL™ 4.0 SF15). The PedsQL™ 4.0 SF15 Questionnaires was completed by all the participants. It is a comprehensive and widely used patient-reported outcome survey designed to measure health-related quality of life in healthy children and adolescents. It was presented for each of the 4 domains of the SF-15 (physical functioning, emotional functioning, social functioning, and school functioning), the psychosocial health summary (emotional, social, and school functioning domains), physical health summary and the Total Score. Total scores as well as each of the subscale scores are transformed on a scale from 0 to 100. Higher scores in each case indicate better HRQOL. A positive change from baseline indicates improvement.
Time Frame: Baseline (Day 1); Weeks 8, FU-12, and FU-24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 21
score on a scale
  Physical Functioning; Baseline | 90.7 (13.81)
  Physical Functioning; Change at Week 8 | -2.6 (10.20)
  Physical Functioning; Change at FU-12 | -3.3 (11.87)
  Physical Functioning; Change at FU-24 | -3.5 (12.72)
  Emotional Functioning; Baseline | 73.2 (20.07)
  Emotional Functioning; Change at Week 8 | 4.8 (10.63)
  Emotional Functioning; Change at FU-12 | 1.8 (19.78)
  Emotional Functioning; Change at FU-24 | 3.0 (15.64)
  Social Functioning; Baseline | 93.3 (12.53)
  Social Functioning; Change at Week 8: number analyzed (Participants) | 20
  Social Functioning; Change at Week 8 | 0.4 (9.16)
  Social Functioning; Change at FU-12 | -2.0 (10.17)
  Social Functioning; Change at FU-24 | -0.8 (8.70)
  School Functioning; Baseline | 75.0 (24.58)
  School Functioning; Change at Week 8 | 5.2 (17.97)
  School Functioning; Change at FU-12 | 0.4 (12.21)
  School Functioning; Change at FU-24 | 1.6 (11.06)
  Physical Health; Baseline | 90.7 (13.81)
  Physical Health; Change at Week 8 | -2.6 (10.20)
  Physical Health; Change at FU-12 | -3.3 (11.87)
  Physical Health, Change at FU-24 | -3.5 (12.72)
  Psychosocial Health; Baseline | 79.8 (14.16)
  Psychosocial Health; Change at Week 8 | 3.8 (7.47)
  Psychosocial Health; Change at FU-12 | 0.2 (9.74)
  Psychosocial Health; Change at FU-24 | 1.4 (8.81)
  Total Score; Baseline | 83.4 (12.40)
  Total Score; Change at Week 8 | 1.7 (5.30)
  Total Score; Change at FU-12 | -1.0 (8.83)
  Total Score; Change at FU-24 | -0.2 (8.58)

24. Secondary Outcome: Change From Baseline in Neuropsychiatric Assessments as Completed by Parent/Legal Guardian
Description: Neuropsychiatric safety assessment was done using the Pediatric Quality of Life (PedsQL™ 4.0 SF15). The PedsQL™ 4.0 SF15 Questionnaires was completed by the parent/ legal guardian of the participants. It is a comprehensive and widely used patient-reported outcome survey designed to measure health-related quality of life in healthy children and adolescents. It is presented for each of the 4 domains of the SF-15 (physical functioning, emotional functioning, social functioning, and school functioning), the psychosocial health summary (emotional, social, and school functioning domains), physical health summary and the Total Score. Total scores as well as each of the subscale scores are transformed on a scale from 0 to 100. Higher scores in each case indicate better HRQOL. A positive change from baseline indicates improvement.
Time Frame: Baseline (Day 1); Weeks 8, FU-12, and FU-24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOF/VEL/VOX FDC
Number analyzed (Participants) | 20
score on a scale
  Physical Functioning; Baseline | 85.3 (22.56)
  Physical Functioning; Change at Week 8 | 3.5 (20.97)
  Physical Functioning; Change at FU-12: number analyzed (Participants) | 19
  Physical Functioning; Change at FU-12 | 2.1 (20.90)
  Physical Functioning; Change at FU-24 | 4.0 (19.97)
  Emotional Functioning; Baseline | 73.4 (18.57)
  Emotional Functioning; Change at Week 8 | 7.8 (18.57)
  Emotional Functioning; Change at FU-12: number analyzed (Participants) | 19
  Emotional Functioning; Change at FU-12 | 6.6 (14.50)
  Emotional Functioning; Change at FU-24 | 4.7 (12.80)
  Social Functioning; Baseline | 85.8 (18.36)
  Social Functioning; Change at Week 8 | 1.3 (21.84)
  Social Functioning; Change at FU-12: number analyzed (Participants) | 19
  Social Functioning; Change at FU-12 | 6.1 (18.39)
  Social Functioning; Change at FU-24 | 2.1 (21.27)
  School Functioning; Baseline | 72.5 (27.59)
  School Functioning; Change at Week 8 | 0.4 (23.64)
  School Functioning; Change at FU-12: number analyzed (Participants) | 19
  School Functioning; Change at FU-12 | 3.9 (22.80)
  School Functioning; Change at FU-24 | 3.8 (20.50)
  Physical Health; Baseline | 85.3 (22.56)
  Physical Health; Change at Week 8 | 3.5 (20.97)
  Physical Health; Change at FU-12: number analyzed (Participants) | 19
  Physical Health; Change at FU-12 | 2.1 (20.90)
  Physical Health, Change at FU-24 | 4.0 (19.97)
  Psychosocial Health; Baseline | 76.8 (17.34)
  Psychosocial Health; Change at Week 8 | 3.7 (17.39)
  Psychosocial Health; Change at FU-12: number analyzed (Participants) | 19
  Psychosocial Health; Change at FU-12 | 5.7 (15.31)
  Psychosocial Health; Change at FU-24 | 3.7 (15.52)
  Total Score; Baseline | 79.7 (15.40)
  Total Score; Change at Week 8 | 3.6 (15.84)
  Total Score; Change at FU-12: number analyzed (Participants) | 19
  Total Score; Change at FU-12 | 4.5 (14.37)
  Total Score; Change at FU-24 | 3.8 (14.89)

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date (maximum: 8 Weeks) plus 30 days
Description: The Safety Analysis Set included participants received at least 1 dose of study drug.
Arm/Group | SOF/VEL/VOX FDC
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX FDC (N=21)
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX FDC (N=21)
Abdominal pain (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 2
Fatigue (General disorders) | 3
Rhinitis (Infections and infestations) | 3
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03820258/SAP_000.pdf
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03820258/Prot_001.pdf